CLINICAL TRIAL: NCT04641780
Title: "Brexpiprazole (Rexulti™) Safety and Efficacy Among Filipino Patients (RAISE) - A Post Marketing Surveillance Program"
Acronym: RAISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Otsuka Pharmaceutical, Inc., Philippines (Industry)
Responsible Party: Sponsor
Other Study IDs: 331-414-00243
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia; Major Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rexulti Tablets: Target is 300 patients in the Philippines diagnosed with Schizophrenia and Major Depressive Disorder
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — For the treatment of schizophrenia, the recommended starting dosage for Rexulti™ is 1 mg once daily on Days 1 to 4, taken orally with or without food. The recommended target Rexulti™ dosage is 2 mg to 4 mg once daily. Titrate to 2 mg once daily on Day 5 through Day 7, then to 4 mg on Day 8 based on the patient's clinical response and tolerability. The maximum recommended daily dosage is 4 mg.
  The recommended starting dosage for Rexulti™ as adjunctive therapy for MDD is 0.5 mg or 1 mg once daily, taken orally with or without food. Titrate to 1 mg once daily, then up to the target dosage of 2 mg once daily. Dosage increases should occur at weekly intervals based on the patient's clinical response and tolerability. The maximum recommended daily dosage is 3 mg. It must be periodically reassess to determine the continued need and appropriate dosage for treatment.
  Other Names: Rexulti

SUMMARY:
The objective of this post marketing surveillance is to further gather local data on the safety and efficacy of Brexpiprazole (RexultiTM) Film-coated Tablet in the treatment of schizophrenia and adjunctive therapy of Major Depressive Disorder.

DETAILED DESCRIPTION:
DESIGN OF THE PMS:

This is a post marketing surveillance of 8 weeks duration, on 300 male or female patients diagnosed to have schizophrenia and MDD in the Philippines.

PROCEDURES:

Based on his clinical decision, the attending physician will enroll patients with schizophrenia and MDD to the program. The attending physician will explain to the patient or his legal guardian the purpose of the PMS and will obtain the patient or legal guardian's consent that Brexpiprazole (Rexulti) Film-coated Tablet will be administered.

Data on the safety aspects of Brexpiprazole (Rexulti) Film-coated Tablet will be collected in terms of adverse events. Efficacy will be measured using the Clinical Global Impression (CGI) Scale (Severity and Improvement).

Assessments will be done upon initiation, (Baseline visit), 4 weeks later (Visit 2), until completion of the study week 8 (Study Completion). Demographic information and vital signs will be collected.

DOSAGE AND ADMINISTRATION:

For the treatment of schizophrenia, the recommended starting dosage for Brexpiprazole (Rexulti™) is 1 mg once daily on Days 1 to 4, taken orally with or without food. The recommended target dosage is 2 mg to 4 mg once daily. Titrate to 2 mg once daily on Day 5 through Day 7, then to 4 mg on Day 8 based on the patient's clinical response and tolerability. The maximum recommended daily dosage is 4 mg.

The recommended starting dosage as adjunctive therapy for MDD is 0.5 mg or 1 mg once daily, taken orally with or without food. Titrate to 1 mg once daily, then up to the target dosage of 2 mg once daily. Dosage increases should occur at weekly intervals based on the patient's clinical response and tolerability. The maximum recommended daily dosage is 3 mg. It must be periodically reassess to determine the continued need and appropriate dosage for treatment.

For patients with moderate to severe hepatic impairment (Child-Pugh score ≥7), the maximum recommended dosage is 2 mg once daily for patients with MDD, and 3 mg once daily for patients with schizophrenia.

For patients with moderate, severe or end-stage renal impairment (creatinine clearance CLcr<60 mL/minute), the maximum recommended dosage is 2 mg once daily for patients with MDD and 3 mg once daily for patients with schizophrenia.

STATISTICAL ANALYSIS:

Analysis of data will be limited to descriptive statistics only. Safety will be evaluated based on the reported AEs per assessment. Efficacy will be evaluated using the Clinical Global Impression-Severity (CGI-S) and Clinical Global Impression-Improvement (CGI-I) Scales to monitor severity and improvement from mean baseline score (before initial dose) up to the last assessment (Week 8 - Study Completion).

ELIGIBILITY:
Inclusion Criteria:

* A total of 300 subjects will be included in the trial
* Adults (18 years old and above)
* Male and Female

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 patients in the Philippines diagnosed with Schizophrenia and Major Depressive Disorder
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-08-17 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Safety assessment of patients with Schizophrenia and Major Depressive Disorder | 8 weeks treatment duration
  Safety of Brexpiprazole (Rexulti™) Film-coated Tablet will be evaluated based on the reported AE's per assessment.

SECONDARY OUTCOMES:
Efficacy assessment of patients with Schizophrenia and Major Depressive Disorder using Clinical Global Impression (CGI) Scale | 8 weeks treatment duration
  Efficacy of Brexpiprazole (Rexulti™) Film-coated Tablet will be evaluated using the Clinical Global Impression (CGI) Scale:
  CGI - Severity
  * Numbers and proportions of responders (defined as patients with CGI severity (CGI-S) score of 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill patients) CGI - Improvement
  * Numbers and proportions of responders (defined as patients with CGI improvement (CGI-I) score of 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), 7 (very much worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Otsuka (Philippines) Pharmaceutical Inc., Makati City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT04641780/Prot_000.pdf